CLINICAL TRIAL: NCT07149779
Title: Effect of Calisthenic Exercises Applied To Kickboxing Players on Strength Parameters
Brief Title: Effect of Calisthenic Exercises on Strength Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şükran İRİBALCI (Other)
Responsible Party: Sponsor-Investigator, Şükran İRİBALCI, Assoc. Prof. Dr. Şükran İRİBALCI, Selcuk University
Organization: Selcuk University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SelcukU-SBF-Şİ-01
Record Dates: First submitted 2025-08-09; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: The Effect of 8 Weeks of Calisthenic Exercises on Strength Parameters in Healthy Athletes Who Exercise Regularly
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A total of 20 kickboxers between the ages of 20-26, healthy, and actively involved in this branch for at least 4 years participated in the study. The volunteers participating in the study were randomly divided into two groups as the study and control groups. The study group applied calisthenic strength exercises in addition to routine kickboxing technical training for 8 weeks and 3 days a week, while the control group continued only their weekly routine kickboxing training without applying any strength training. Static strength performance (grip-leg-back), dynamic strength performance (1RM bench press and 1RM barbel squat), 30-second push-ups and 30-second sit-ups tests were applied to the athletes participating in the study before and after the 8-week training.

SUMMARY:
This study was conducted to investigate the effects of a calisthenic exercise program on static/dynamic strength and muscular endurance in young male kickboxers. Methods: A total of 20 kickboxers between the ages of 20-26, healthy, and actively involved in this branch for at least 4 years participated in the study. The volunteers participating in the study were randomly divided into two groups as the study and control groups. The study group applied calisthenic strength exercises in addition to routine kickboxing technical training for 8 weeks and 3 days a week, while the control group continued only their weekly routine kickboxing training without applying any strength training. Static strength performance (grip-leg-back), dynamic strength performance (1RM bench press and 1RM barbel squat), 30-second push-ups and 30-second sit-ups tests were applied to the athletes participating in the study before and after the 8-week training. SPSS 25.0 and JASP statistical package programs were used in the evaluation of the data obtained in the study and the significance level was accepted as 0.05.

DETAILED DESCRIPTION:
Methods:

Study design and participants:

Twenty male kickboxers, aged 20-26, who regularly train and are licensed, participated in the study. After the volunteers who participated in the study were informed about the test protocols, measurements and the general study, they were randomly divided into two groups as the study and control groups. The study group applied calisthenic strength exercises for 8 weeks and 3 days a week in addition to their regular kickboxing training, while the control group continued only their weekly routine kickboxing training. Measurements were made for 3 days with 24-hour intervals so that the physiological effects of the applied tests would not affect other tests. All data obtained from the control and training groups before and after the study were compared and examined.

Data Collection Determination of height and body weight: Before and after the eight-week planned training program, the height and body weight of all participants were determined with an Oncomed brand SC-105 model 0.1 kg precision measuring device and the body mass index (BMI) value was calculated.

30-second push-up test: After the subjects took a position on the floor mat, they were asked to lower their bodies until their elbows reached 90 degrees, with their arms open at shoulder width, elbows straight and tense, without touching the ground and without creating a concave waist, and then return to the starting position after approaching the ground. The number of regular push-ups performed for 30 seconds was recorded.

30-second sit-up test: After the subjects lay on their backs on a mat laid on the floor, their arms were joined on their chests and their knees were at a 45° angle. The subjects were asked to lift their bodies 90° off the ground and touch the ground again in the starting position. The number of regular sit-ups performed for 30 seconds was recorded.

Static strength measurement test: A dynamometer was used to determine the grip, back and leg strength of the subjects.

Dynamic strength measurement test: The maximal weight that all participants in the study could lift at one time was determined with the 1 repetition maximal (1RM) method of the bench press movement, one of the basic exercises for the upper extremity, and the barbell squat movement, which is considered a basic exercise for the lower extremity.

Calisthenic Training Program:

The athletes in the training group of the study were included in a calisthenic training program consisting of burpees, push-ups, sit-ups, bench dips, jumping jacks, jumping squats, mountain climbers, straight and side plank movements in addition to regular kickboxing training. The calisthenic training program was applied to the athletes for 8 weeks, 3 days a week, with each movement lasting 30-60 seconds (starting with 30 seconds and increasing by 10 seconds every two weeks), 15 seconds between repetitions, and 2 minutes between sets, for a total of 2 sets.

Statistical Analysis SPSS 25.0 and JASP statistical package programs were used to evaluate the data obtained in the study, and the significance level was accepted as 0.05. A t-test was applied in independent samples to determine whether there were statistically significant differences between the control and study groups.

ELIGIBILITY:
Inclusion Criteria:

* those who participate in regular training healthy and volunteers

Exclusion Criteria:

* have any injuries
* not participating in regular training

Ages: 20 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Determination of height and body weight | from the beginning of the work until the end of 8 weeks
  All participants were determined with an Oncomed brand SC-105 model 0.1 kg precision measuring device and the body mass index (BMI) value was calculated.
30-second push-up test | from the beginning of the work until the end of 8 weeks
  After the subjects took a position on the floor mat, they were asked to lower their bodies until their elbows reached 90 degrees, with their arms open at shoulder width, elbows straight and tense, without touching the ground and without creating a concave waist, and then return to the starting position after approaching the ground. The number of regular push-ups performed for 30 seconds was recorded.
30-second sit-up test | from the beginning of the work until the end of 8 weeks
  After the subjects lay on their backs on a mat laid on the floor, their arms were joined on their chests and their knees were at a 45° angle. The subjects were asked to lift their bodies 90° off the ground and touch the ground again in the starting position. The number of regular sit-ups performed for 30 seconds was recorded.
Static strength measurement test | from the beginning of the work until the end of 8 weeks
  A dynamometer was used to determine the grip, back and leg strength of the subjects.
Dynamic strength measurement test | from the beginning of the work until the end of 8 weeks
  The maximal weight that all participants in the study could lift at one time was determined with the 1 repetition maximal (1RM) method of the bench press movement, one of the basic exercises for the upper extremity, and the barbell squat movement, which is considered a basic exercise for the lower extremity.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk university, Konya, Turkey (Türkiye)